CLINICAL TRIAL: NCT03125421
Title: A Nursing Strategy to Prevent Pressure Sores in the Prone Position in ARDS Patients. A Multicenter Controlled Prospective Stepped Wedge Trial
Brief Title: Prevention of Pressure Sores in the Prone Position in ARDS Patients
Acronym: PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL17_0039
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pressure Sores
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control period (Other): standard preventive methods of pressure sores in each center
  Interventions: Procedure: standard preventive methods of pressure sores
- experimental period (Experimental): experimental multifaceted preventive methods of pressure sores
  Interventions: Procedure: experimental multifaceted preventive methods of pressure sores

INTERVENTIONS:
Procedure: standard preventive methods of pressure sores — During the control period, the following specific methods to prevent pressure sores in the prone position (in ARDS patients mechanically ventilated via tracheal route) will be these ongoing in each center and involve the following components: lower eyelid and ocular protection by any method, inclination of the body from the horizontal position, intermittent head mobilization to the right or to the left, and no use of specific device to prevent pressures sores at the head and/or thorax, and/or knees, and/or feet.
  The following nonspecific methods to prevent pressures sores will be performed at the discretion of each center according to its usual practice: mattress, upper eyelid protection, main devices securely fasten, arms position, abdomen supported or not, mouth care, enteral nutrition continued in the prone position, skin protection and/or massage.
  Arms: control period
Procedure: experimental multifaceted preventive methods of pressure sores — During the experimental period, the following specific methods to prevent pressure sores in the prone position (in ARDS patients mechanically ventilated via tracheal route) will be systematically applied: lower eyelid protection by horizontal strap, ocular protection by methylcellulose, 15° inclination of the body from the horizontal position, intermittent head mobilization to the right or to the left every four hours, and use of specific device to prevent pressures sores at the head, thorax, knees, and feet.
  The following nonspecific methods to prevent pressures sores will be applied as in the control period described above except for the following: the abdomen will not be supported and the skin will not be protected.
  Arms: experimental period

SUMMARY:
A nursing strategy to prevent pressure sores in the prone position in Acute Respiratory Distress Syndrome (ARDS) patients. A multicenter controlled prospective stepped wedge trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more in age
* staying in Intensive Care Unit (ICU)
* Intubated
* mechanically ventilated
* severe ARDS defined as arterial Pressure in Oxygen (PaO2)/ Oxygen Inspired Fraction (FIO2) < 150 mmHg with positive end-expiratory pressure (PEEP) ≥ 5 cmH2O and FIO2 ≥ 0.60
* prone positioning indicated by the clinician in charge
* weight < 140 kgs
* agreement to participate obtained from the confidence person of the patient
* affiliated to social protection insurance

Exclusion Criteria:

* contra-indication to the prone positioning
* prone positioning before inclusion
* person under legal protection
* pregnancy
* weight > 140 kg
* tracheotomy
* extracorporeal membrane oxygenation (ECMO)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
number of patients with a new pressure sore of any stage in any predetermined location | day 7 after inclusion
  New pressure sores are validated by the independent committee (2 persons) in charge of the analysis of the pictures performed in the patients. The whole body is pictured in 3 parts and specific locations will be analyzed, which are forehead, nose, eyes, chin, jaw, lips, thorax, breast, knee, iliac crest, foot extension area, and external genitalia in man. For each location a four-stage severity score of the pressure sore is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Gay, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hopital Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gay L, Huot L, Yonis H, Valera S, Hraeich S, Matthieu D, Gacouin A, Ouisse C, Reignier J, Massard A, Quenot JP, Revol C, Robine A, Guillemault O, Bourdin G, Robert A, Lacherade JC, Perarder C, Badet M, Baboi L, Rabilloud M, Decullier E, Montagne E, Girard R, Arcuset C, Mevel J, de Montigny AM, Guerin C. A Bundle of Interventions to Prevent Pressure Ulcers During Prone Position in Adult Patients With Acute Respiratory Distress Syndrome: Results of a French Stepped-Wedge Randomized Controlled Trial. Nurs Crit Care. 2025 Jul;30(4):e70084. doi: 10.1111/nicc.70084. PMID 40509643